CLINICAL TRIAL: NCT02222168
Title: Open, Randomised, Two-way Crossover Study to Assess the Effect of a High Fat, High Caloric Meal on the Pharmacokinetics of BI 409306, Followed by a Fixed Sequence Period to Investigate the Pharmacokinetics of BI 409306 After a Single Oral Dose Given at Bed Time in Healthy Male and Female Volunteers
Brief Title: Pharmacokinetics of BI 409306 After a High Fat, High Caloric Meal and After a Single Oral Dose Given at Bed Time in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1289.22; 2014-001934-28 (EudraCT Number: EudraCT)
Record Dates: First submitted 2014-08-20; First posted 2014-08-21 (Estimated); Results first posted 2024-03-07 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Healthy
MeSH Terms: interventions — BI 409306

ARMS (3):
- BI 409306 fasted (Experimental): Single dose 25 mg BI 409306 film-coated tablet, oral administration with 240 ml water in the morning under fasted condition.
  Interventions: Drug: BI 409306
- BI 409306 fed (Experimental): Single dose 25 mg BI 409306 film-coated tablet, oral administration with 240 ml water in the morning under fed condition.
  Interventions: Drug: BI 409306
- BI 409306 at bed-time (Experimental): Single dose 25 mg BI 409306 film-coated tablet, oral administration with 240 ml water at bed-time.
  Interventions: Drug: BI 409306

INTERVENTIONS:
Drug: BI 409306 — film-coated tablet

SUMMARY:
To evaluate the effect of food on the pharmacokinetics of BI 409306 and to investigate the pharmacokinetics of BI 409306 when given at bed time.

ELIGIBILITY:
Inclusion criteria:

1. Healthy male and female volunteers
2. Age 18 (incl.) to 50 (incl.) years
3. Body mass index (BMI) range: 18.5 (incl.) to 29.9 (incl.) kg/m2

Exclusion criteria:

1. Any evidence of a clinically relevant concomitant disease
2. Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
4. Surgery of the gastrointestinal tract (except appendectomy)
5. Diseases of the central nervous system (including but not limited to any kind of seizures, stroke or psychiatric disorders)
6. History or evidence of relevant orthostatic reaction, fainting spells or blackouts, occurrence of syncopes, brady- or tachycardia in the anamnesis.
7. Positive pregnancy test
8. No adequate contraception during the study and until 1 month of study completion, i.e. intrauterine device (IUD), sexual abstinence (for at least 1 month prior to enrolment), or surgical sterilisation (incl. hysterectomy). Females, who are not surgically sterile will be asked to additionally use barrier contraception methods (e.g. condom, diaphragm with spermicide)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2014-09-04 (Actual); Primary Completion 2014-10-31 (Actual); Study Completion 2014-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1289.22.1 Boehringer Ingelheim Investigational Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization). For more details refer to: https:// www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eighteen healthy subjects were entered and treated and completed the planned observation time. All 18 subjects received study medication (open-label) under fasted (Treatment A) and fed (Treatment B) conditions in a two-way crossover fashion followed by a fixed sequence administered at bed time (Treatment C).
Pre-assignment Details: All subjects were screened for eligibility to participate in the trial. Subjects attended specialist sites which would then ensure that the subject met all strictly implemented inclusion/exclusion criteria. Subjects were not to be randomised to trial treatment if any one of the specific entry criteria were violated.
Groups:
- BI 409306 Fasted/Fed/Bed Time: Single oral dose of 25 milligram (mg) BI 409306 film-coated tablet, with 240 millilitre (ml) water in the morning under fasted then under fed condition and last administered at bed-time with a washout period of at least 3 days between the administrations.
- BI 409306 Fed/Fasted/Bed Time: Single oral dose of 25 mg BI 409306 film-coated tablet, with 240 ml water in the morning under fed then under fast condition and last administered at bed-time with a washout period of at least 3 days between the administrations.
Period: Period 1 (Fasted or Fed)
Arm/Group | BI 409306 Fasted/Fed/Bed Time | BI 409306 Fed/Fasted/Bed Time
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0
Period: Period 2 (Fasted or Fed)
Arm/Group | BI 409306 Fasted/Fed/Bed Time | BI 409306 Fed/Fasted/Bed Time
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0
Period: Period 3 (Bed-time)
Arm/Group | BI 409306 Fasted/Fed/Bed Time | BI 409306 Fed/Fasted/Bed Time
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The treated set (TS): This set included all subjects who received at least one dose of trial medication. It was used for the analysis of safety, demographic data, baseline characteristics, and disposition. The TS included all 18 subjects.
Groups:
- BI 409306 Fasted/Fed/Bed Time: Single oral dose of 25 mg BI 409306 film-coated tablet, with 240 ml water in the morning under fasted then under fed condition and last administered at bed-time with a washout period of at least 3 days between the administrations.
- Total: Total of all reporting groups
Arm/Group | BI 409306 Fasted/Fed/Bed Time | BI 409306 Fed/Fasted/Bed Time | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.2 (5.4) | 44.3 (9.1) | 37.3 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 5 | 6 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 9 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Measured Concentration of BI 409306 in Plasma (Cmax)
Description: Cmax is the maximum measured concentration of BI 409306 in plasma. More detailed time frame information: 1 hour (h) before administration of BI 409306 and 0:10, 0:20, 0:30, 0:45, 1:00, 1:30, 2:00, 2:30, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 14:00, 24:00 h after administration of BI 409306 at treatment A/B; 1h before administration of BI 409306 and 0:10, 0:20, 0:30, 0:45, 1:00, 1:30, 2:00, 2:30, 4:00, 6:00, 8:00, 10:00, 12:00, 14:00, 24:00 h after administration of BI 409306 at treatment C
Time Frame: Treatment A/B: -1:00, 0:10, 0:20, 0:30, 0:45, 1:00, 1:30, 2:00, 2:30, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 14:00, 24:00h; treatment C: -1:00, 0:10, 0:20, 0:30, 0:45, 1:00, 1:30, 2:00, 2:30, 4:00, 6:00, 8:00, 10:00, 12:00, 14:00, 24:00h
Population: The Pharmacokinetic set (PKS): This set included all treated subjects who provided at least one observation for at least one primary endpoint without important protocol violations with respect to the statistical evaluation of PK endpoints. All 18 subjects were included in the PKS.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomole per litre
Arm/Group | BI 409306 Fasted | BI 409306 Fed | BI 409306 at Bed-time
Number analyzed (Participants) | 18 | 18 | 18
Nanomole per litre | 183 (118) | 175 (69.5) | 150 (119)
Statistical Analysis 1: Comparison: BI 409306 Fasted vs BI 409306 Fed; No formal hypothesis was tested; Test type: Other — The statistical model used for the analysis of the endpoint comparing 'BI 409306 fasted' against 'BI 409306 fed' was an Analysis of Variance (ANOVA ) model on the logarithmic scale.This model included effects accounting for the following sources of variation: 'sequence', 'subjects within sequences', 'period' and'treatment'. The effect 'subjects within sequences' was considered as random, whereas the other effects were considered as fixed; Ratio (Fed/Fasted) = 95.90, 90% CI 2-sided [72.593 to 126.682], Standard Error of Mean 50.7 — The estimated parameter was the adjusted geometric mean ratios [%] of BI 409306: fed (numerator), fasted (denominator). The standard deviation is the intra-individual geometric coefficient of variation [%]
Statistical Analysis 2: Comparison: BI 409306 Fasted vs BI 409306 at Bed-time; No formal hypothesis was tested; Test type: Other — The statistical model used for the analysis of the endpoint comparing 'BI 409306 fasted' against 'BI 409306 at bed-time' was an Analysis of Variance (ANOVA ) model on the logarithmic scale. This model included effects accounting for the following sources of variation: 'subject' and 'treatment'. The effect 'subject' was considered as random, whereas the effect treatment was considered as fixed; Ratio (Bed time/Fasted) = 82.13, 90% CI 2-sided [66.370 to 101.639], Standard Error of Mean 38.0 — The estimated parameter was the adjusted geometric mean ratios [%] of BI 409306: at bed time (numerator), fasted (denominator). The standard deviation is the intra-individual geometric coefficient of variation [%]

2. Primary Outcome: Area Under the Concentration-time Curve of BI 409306 in Plasma From Time 0 to Time of Last Quantifiable Data Point (AUC0-tz)
Description: AUC0-tz is the area under the concentration-time curve of the BI 409306 in plasma from time 0 to time of last quantifiable data point.
  More detailed time frame information: 1 hour (h) before administration of BI 409306 and 0:10, 0:20, 0:30, 0:45, 1:00, 1:30, 2:00, 2:30, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 14:00, 24:00 h after administration of BI 409306 at treatment A/B; 1h before administration of BI 409306 and 0:10, 0:20, 0:30, 0:45, 1:00, 1:30, 2:00, 2:30, 4:00, 6:00, 8:00, 10:00, 12:00, 14:00, 24:00 h after administration of BI 409306 at treatment C
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour times nanomole per litre
Arm/Group | BI 409306 Fasted | BI 409306 Fed | BI 409306 at Bed-time
Number analyzed (Participants) | 18 | 18 | 18
Hour times nanomole per litre | 273 (118) | 293 (96.4) | 259 (117)
Statistical Analysis 1: Comparison: BI 409306 Fasted vs BI 409306 Fed; No formal hypothesis was tested; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio (Fed/Fasted) = 107.41, 90% CI 2-sided [96.697 to 119.318], Standard Error of Mean 18.2 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: BI 409306 Fasted vs BI 409306 at Bed-time; No formal hypothesis was tested; Test type: Other — [test comment as in outcome 1, analysis 2]; Ratio (Bed time/Fasted) = 94.88, 90% CI 2-sided [85.028 to 105.875], Standard Error of Mean 19.1 — [estimate comment as in outcome 1, analysis 2]

3. Secondary Outcome: Area Under the Concentration-time Curve of BI 409306 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-infinity)
Description: AUC0-infinity is the area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity.
  More detailed time frame information: 1 hour (h) before administration of BI 409306 and 0:10, 0:20, 0:30, 0:45, 1:00, 1:30, 2:00, 2:30, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 14:00, 24:00 h after administration of BI 409306 at treatment A/B; 1h before administration of BI 409306 and 0:10, 0:20, 0:30, 0:45, 1:00, 1:30, 2:00, 2:30, 4:00, 6:00, 8:00, 10:00, 12:00, 14:00, 24:00 h after administration of BI 409306 at treatment C.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour times nanomole per litre
Arm/Group | BI 409306 Fasted | BI 409306 Fed | BI 409306 at Bed-time
Number analyzed (Participants) | 18 | 18 | 18
Hour times nanomole per litre | 273 (118) | 293 (96.3) | 259 (116)
Statistical Analysis 1: Comparison: BI 409306 Fasted vs BI 409306 Fed; No formal hypothesis was tested; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio (Fed/Fasted) = 107.41, 90% CI 2-sided [96.709 to 119.301], Standard Error of Mean 18.2 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: BI 409306 Fasted vs BI 409306 at Bed-time; No formal hypothesis was tested; Test type: Other — [test comment as in outcome 1, analysis 2]; Ratio (Bed time/Fasted) = 94.92, 90% CI 2-sided [85.061 to 105.921], Standard Error of Mean 19.1 — [estimate comment as in outcome 1, analysis 2]

ADVERSE EVENTS:
Time Frame: From first administration of BI 409306 up to 24 hours thereafter for each treatment period.
Arm/Group | BI 409306 Fasted | BI 409306 Fed | BI 409306 at Bed-time
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 1/18 | 4/18 | 1/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 409306 Fasted (N=18) | BI 409306 Fed (N=18) | BI 409306 at Bed-time (N=18)
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Feeling hot (General disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 2 | 0
Headache (Nervous system disorders) | 0 | 1 | 1
Bladder discomfort (Renal and urinary disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.